CLINICAL TRIAL: NCT06729008
Title: Effect of Diabetes-Specific Nutrition Formula on the Metabolic Parameters of Filipino Adults with Metabolic Syndrome: a Randomized Crossover Trial
Brief Title: Effect of Diabetes-Specific Nutrition Formula on the Metabolic Parameters of Filipino Adults with Metabolic Syndrome
Acronym: DSNFMETSPH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's Medical Center, Philippines (Other)
Responsible Party: Principal Investigator, Angelica Marie Real, Principal Investigator, St. Luke's Medical Center, Philippines
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CDTEDDSNF2025
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Diabetes-Specific Nutrition Formula; Philippines
MeSH Terms: conditions — Metabolic Syndrome | interventions — Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DSNF + MNT (Experimental)
  Interventions: Dietary Supplement: Diabetes-specific nutrition formula (DSNF); Other: Medical Nutrition Therapy
- MNT (Active Comparator)
  Interventions: Other: Medical Nutrition Therapy

INTERVENTIONS:
Dietary Supplement: Diabetes-specific nutrition formula (DSNF) — The diabetes-specific nutrition formula to be used in this study will be Glucerna (Abbott Laboratories). It features an advanced blend of low-glycemic carbohydrates for steady energy release, a dual fiber blend to support digestive health, and a unique lipid blend free from trans fats, cholesterol, and low in saturated fat. Additionally, Glucerna is enriched with 4x more inositol and high levels of trivalent chromium, which contribute to maintaining normal blood glucose levels. It provides 28 essential vitamins and minerals, is low in lactose, and gluten-free, making it a suitable option for various dietary needs. 5 scoops will be mixed in 200 mL of water, and this amounts to 228 calories, with 30.01g of carbohydrates, 10.16g of protein, and 8.70g of fat. This will be given twice, as a breakfast replacement and an afternoon snack replacement.
  Arms: DSNF + MNT
Other: Medical Nutrition Therapy — Medical Nutrition Therapy is the standard of care for the management of metabolic syndrome
  Other Names: MNT

SUMMARY:
INTRODUCTION: Metabolic syndrome, a cluster of metabolic abnormalities, is a growing global health concern, particularly in the Asia-Pacific region. The Philippines has seen a significant rise in metabolic syndrome prevalence, linked to lifestyle factors and socioeconomic changes. This condition increases the risk of serious health issues like type 2 diabetes, cardiovascular disease, and mortality. Lifestyle modifications, including dietary interventions, are crucial for managing metabolic syndrome. While dietary recommendations exist, practical challenges hinder their implementation. Diabetes-specific nutrition formulas (DSNFs) offer a convenient and effective solution, especially for individuals with limited cooking skills or knowledge. While DSNFs show promise in managing diabetes, their impact on metabolic syndrome remains unclear. This study aims to investigate the effects of DSNF on the metabolic parameters of Filipino adults with metabolic syndrome.

METHODS: This open-label randomized crossover trial will be conducted at St. Luke's Medical Center Global City. Filipino adults aged 19-65 with metabolic syndrome will be recruited. Participants will be randomized to either a 90-day intervention phase (DSNF) with a 14-day washout period or a 90-day control phase. After the initial phase, participants will cross over to the alternate phase. The primary outcome will be the change in metabolic parameters in the metabolic syndrome criteria (fasting blood sugar, triglycerides, HDL cholesterol, blood pressure, and waist circumference). Secondary outcomes include changes in metabolic parameters related to the metabolic syndrome (glycosylated hemoglobin, total cholesterol, LDL cholesterol, body weight, BMI, body composition), and safety and tolerability of the treatments. Participants will be monitored through regular follow-up visits, daily food diaries, and subjective assessments. Data will be analyzed using appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

1. An employee of St. Luke's Medical Center Global City for at least 1 year
2. Of Filipino descent
3. Aged 19-65 years
4. Diagnosed with metabolic syndrome74 for at least 3 months, one of the criteria must include central obesity (WC of ≥90cm in Asian men, ≥80cm in Asian women)

   a. If being treated with a stable dose of medications for metabolic syndrome for ≥ 1 month, must only be among the following: i. Oral hypoglycemic agents (OHAs) (drugs permitted include Metformin, Sulfonylureas, Thiazolidinedione, Dipeptidyl Peptidase-IV Inhibitors, Glucagon-Like Peptide-1 Agonists) ii. Anti-hypertensive medications (drugs permitted include Angiotensin-converting enzyme (ACE) inhibitors, Angiotensin II receptor blockers, Calcium Channel Blockers) iii. Medications treating dyslipidemia (drugs permitted include Statins, Fibrates, Ezetimibe)
5. BMI of 23 kg/m2 or more
6. Willingness to adhere to study protocol

Exclusion Criteria:

1. Serious illness requiring medical attention within past year (active malignancy, HIV/AIDS, cardiovascular, respiratory, renal, or hepatic diseases)
2. Use of medications affecting plasma glucose within 3 months (corticosteroids, diuretics, beta-blockers, antipsychotics, and HIV medications)
3. Insulin use
4. Severe hypoglycemia or hyperglycemia requiring hospitalization within past year
5. Surgery or hospitalization within past 2-3 months
6. Anemia and/or blood transfusion within the last 3 months
7. History of gastrointestinal disease/surgery affecting product consumption/absorption (inflammatory bowel disease/bowel resection, another specifies gastroparesis, malabsorption, bariatric surgery, short bowel syndrome)
8. Use of other diabetes-specific formulas prior to this study
9. Use of nutritional food supplements or multivitamin supplements (specifically calcium/vitamin D supplements and B complex syrups) within 15 days before study initiation
10. Psychiatric disorder impairing study adherence (eating disorders, severe dementia, delirium, significant neurological/psychiatric disorder)
11. Pregnancy/ lactation
12. Allergy/intolerance to study product components (INGREDIENTS : Maltodextrin, VEGETABLE OIL (high oleic sunflower oil, soy oil), calcium caseinate, sucromalt, isolated soy protein, maltitol, milk protein concentrate (cow's milk), MINERALS (potassium chloride, magnesium sulfate, calcium carbonate, potassium citrate, sodium phosphate, sodium chloride, magnesium phosphate, sodium citrate, potassium hydroxide, zinc sulfate, ferrous sulfate, manganese sulfate, copper sulfate, chromium chloride, potassium iodide, sodium molybdate, sodium selenite), fructose, fructo-oligosaccharides, isomaltulose, myo-inositol, oat fiber, flavoring, emulsifier (carboxymethyl cellulose), choline chloride, emulsifier (soy lecithin), stabiliser (xanthan gum), VITAMINS (ascorbyl palmitate, ascorbic acid, Vitamin E, niacinamide, calcium d-pantothenate, pyridoxine hydrochloride, thiamin chloride hydrochloride, riboflavin, Vitamin A palmitate, folic acid, phylloquinone, d-biotin, cholecalciferol, cyanocobalamin), taurine, L-carnitine, mixed tocopherols. Contains permitted flavouring substance. Contains stabilisers and emulsifiers as permitted food conditioners.)
13. Weight loss/gain ≥ 5 kg within 6 weeks of starting the study
14. Planning to start any form of calorie-restricted diet
15. Alcoholism/substance use

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
change from baseline to post-intervention in fasting blood sugar | 3 months
  The primary outcome measure of this study is the change from baseline to post-intervention in the following parameter of metabolic syndrome: fasting blood sugar, measured in mg/dL.
change from baseline to post-intervention in HDL cholesterol | 3 months
  The primary outcome measure of this study is the change from baseline to post-intervention in the following parameter of metabolic syndrome: HDL cholesterol, measured in mg/dL.
change from baseline to post-intervention in serum triglycerides | 3 months
  The primary outcome measure of this study is the change from baseline to post-intervention in the following parameter of metabolic syndrome: serum triglycerides, measured in mg/dL.
change from baseline to post-intervention in systolic blood pressure | 3 months
  The primary outcome measure of this study is the change from baseline to post-intervention in the following parameter of metabolic syndrome: systolic blood pressure, measured in mmHg.
change from baseline to post-intervention in diastolic blood pressure | 3 months
  The primary outcome measure of this study is the change from baseline to post-intervention in the following parameter of metabolic syndrome: diastolic blood pressure, measured in mmHg.
change from baseline to post-intervention in waist circumference | 3 months
  The primary outcome measure of this study is the change from baseline to post-intervention in the following parameter of metabolic syndrome: waist circumference, measured in centimeters.

SECONDARY OUTCOMES:
change from baseline to post-intervention in glycosylated hemoglobin | 3 months
  The secondary outcome measures of this study are the change from baseline to post-intervention in the following parameter related to metabolic syndrome: glycosylated hemoglobin, measured as a percentage of total hemoglobin.
change from baseline to post-intervention in LDL cholesterol | 3 months
  The secondary outcome measures of this study are the change from baseline to post-intervention in the following parameter related to metabolic syndrome: LDL cholesterol, measured in mg/dL.
change from baseline to post-intervention in total cholesterol | 3 months
  The secondary outcome measures of this study are the change from baseline to post-intervention in the following parameter related to metabolic syndrome: total cholesterol, measured in mg/dL.
change from baseline to post-intervention in body weight | 3 months
  The secondary outcome measures of this study are the change from baseline to post-intervention in the following parameter related to metabolic syndrome: body weight, measured in kilograms.
change from baseline to post-intervention in body mass index | 3 months
  The secondary outcome measures of this study are the change from baseline to post-intervention in the following parameter related to metabolic syndrome: body mass index, measured in kg/m^2.
Adverse events related to the DSNF | 3 months
  Adverse events related to the DSNF such as diarrhea, constipation, abdominal distension, bloating, nausea, vomiting, and flatulence
Satiety scale | 3 months
  A visual analog scale called the SLIM scale (satiety labeled intensity magnitude scale) will assess participants' subjective feelings of fullness or satiety. This will also be asked daily per meal via Google Forms. The SLIM scale is a vertical line anchored by "greatest imaginable fullness" at one end at 100mm, and "greatest imaginable hunger" at the other at -100mm. Descriptive phrases indicating various hunger and fullness levels are placed along the scale.
DSNF Compliance | 3 months
  Compliance with the DSNF will be determined by reviewing the participants' daily food diary and returned product cans. 1 can contains 35 scoops. The compliance percentage will be calculated as: (number of scoops consumed per day/ number of scoops prescribed per day) * 100. This will also be counterchecked by counting the number of scoops in the returned product cans.
Participants' perception of DSNF | 3 months
  This will be assessed using a 9-point hedonic scale. The 9-point hedonic scale will consist of "dislike extremely", "dislike very much", "dislike moderately", "dislike slightly", "neither like nor dislike", "like slightly", "like moderately", "like very much", and "like extremely". In addition to the hedonic scale, an open-ended question will be included to allow participants to express their thoughts and opinions about the product.

CONTACTS AND LOCATIONS:
Overall Officials: Joy Arabelle C Fontanilla, Doctor of Medicine, Principal Investigator — St. Luke's Medical Center, Philippines; Maria Patricia Deanna D Maningat, Doctor of Medicine, Principal Investigator — St. Luke's Medical Center, Philippines; Sahra May O Paragas, Doctor of Medicine, Principal Investigator — St. Luke's Medical Center, Philippines

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zimmet P, Alberti KG, Shaw J. Global and societal implications of the diabetes epidemic. Nature. 2001 Dec 13;414(6865):782-7. doi: 10.1038/414782a. PMID 11742409
- [Background] International Diabetes Federation. The IDF consensus worldwide definition of the metabolic syndrome. Accessed November 7, 2024. https://idf.org/media/uploads/2023/05/attachments-30.pdf
- [Background] Amihaesei IC, Chelaru L. Metabolic syndrome a widespread threatening condition; risk factors, diagnostic criteria, therapeutic options, prevention and controversies: an overview. Rev Med Chir Soc Med Nat Iasi. 2014 Oct-Dec;118(4):896-900. PMID 25581945
- [Background] Ranasinghe P, Mathangasinghe Y, Jayawardena R, Hills AP, Misra A. Prevalence and trends of metabolic syndrome among adults in the asia-pacific region: a systematic review. BMC Public Health. 2017 Jan 21;17(1):101. doi: 10.1186/s12889-017-4041-1. PMID 28109251